CLINICAL TRIAL: NCT03455517
Title: Activity and Safety of Front-linevenetoclax and Rituximab Association (VeRiTAs) in Young and Fit Patients With Chronic Lymphocytic Leukemia (CLL) and Umutated IGVH and/or Disrupted TP53. A Phase 2 Multicenter Study
Brief Title: Activity and Safety of Front-line Venetoclax and Rituximab in Young and Fit Patients With Chronic Lymphocytic Leukemia
Acronym: VeRitAs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLC1518
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; Umutated IGVH; Disrupted TP53
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — venetoclax; Rituximab

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, interventional, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Veritas (Experimental): * Step 1. All patients: venetoclax 5-weeks dose-titration phase with weekly increases in the dose of venetoclax.
  * Step 2. All patients will receive 6 courses of the VR combination.
  * Step 3. After 6 courses of VR combination:
    3a. Patients with no response will be off treatment; 3b. Patients with clinical response (CR or PR) after 6 courses of VR combination will receive venetoclax as a single agent for 6 months. Then, patients will be observed clinically until disease progression or until month 36.
  Interventions: Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Venetoclax — Venetoclax and rituximab association
Drug: Rituximab — Venetoclax and rituximab association

SUMMARY:
Fludarabine, cyclophosphamide, and rituximab (FCR) is the gold treatment for fit and young patients with Chronic Lymphoid Leukemia (CLL). However, patients with a mutation known as IGVH unmutated and patients with a particular characteristic known as 'disrupted TP53' show an inferior outcome after FCR in terms of survival. Venetoclax as a single agent or combined with rituximab is an effective treatment for relapsed/refractory patients with IGVH unmutated CLL and/or del(17p) and is associated with a high rate of clinical responses.

DETAILED DESCRIPTION:
Fludarabine, cyclophosphamide, and rituximab (FCR) is the gold treatment for fit and young (age ≤65 years) patients with CLL. However, IGVH unmutated patients and patients with disrupted TP53 show an inferior outcome after FCR in terms of PFS and OS. Venetoclax as a single agent or combined with rituximab is an effective treatment for relapsed/refractory patients with IGVH unmutated CLL and/or del(17p) and is associated with a high rate of clinical responses and MRD-negative responses. The achievement of a MRD negative response in CLL is the best treatment endpoint since it is associated with an improved PFS.

In treatment-naive patients with unmutated IGVH and/or disrupted TP53 the venetoclax and rituximab combination could be a more effective regimen than FCR with a 15% increase in the CR rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than18 years and 65 years or less.
* Diagnosis of CLL meeting the IWCLL 2008 criteria.
* Total CIRS <6, creatinine clearance >30 ml/min [Cockcroft-Gault]) and ECOG performance status of 0-1.
* No prior treatment.
* Umutated IGVH and/or disrupted TP53.
* Active disease meeting at least 1 of the following the IWCLL 2008 criteria for treatment requirement.
* Adequate bone marrow function without transfusion <2 weeks of screening as follows: absolute neutrophil count (ANC) ≥1.0 x 109/L (growth factors administration is allowed); platelets ≥30 x 109/L. If thrombocytopenia due to BM involvement, platelets should be ≥ 30 x 109/L; hemoglobin value ≥8.0 g/dl.
* Adequate renal and hepatic function per local reference laboratory reference ranges
* Female patients of childbearing potential and non-sterile male patients must practice at least one of method of birth control with partner(s) beginning with initial treatment administration and continuing to 12 months after the last dose of Rituximab.
* Male patients must agree to refrain from sperm donation, from initial treatment administration until 12 months after the last dose of Rituximab.
* A signed informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

* Any significant concurrent, uncontrolled medical condition or organ system dysfunction and/or laboratory abnormality or psychiatric disease, which, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk or prevent the subject from signing the informed consent form.
* Transformation of CLL to aggressive NHL (Richter's transformation or pro-lymphocytic leukemia).
* History of other malignancies Pregnant or lactating females.
* Inadequate renal function: CrCl <30 mL/min.
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
* Subject is known to be positive for HIV.
* Evidence of other clinically significant uncontrolled condition(s)
* Prior or concomitant fruits and/or specific drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving complete response (CR) | At 15 months from treatment start, which is the end of treatment

SECONDARY OUTCOMES:
Number of patients achieving response | At 15 months from treatment start, which is the end of treatment
  Overall response rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Romana Mauro, Principal Investigator — Università degli Studi di Roma "Sapienza"
Locations (31):
- Italy (31):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Asl Di Asti, Ospedali Riuniti - Presidio Ospedaliero Cardinal G. Massaia - Sc Oncologia, Asti
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - Ao Di Catanzaro "Pugliese-Ciaccio", Presidio Ospedaliero "Ciaccio - de Lellis" - Ematologia, Catanzaro
  - Aou Arcispedale Sant'Anna - Cona (Fe) - Uoc Ematologia E Fisiopatologia Della Coagulazione, Cona
  - Aso S. Croce E Carle - Cuneo - Sc Ematologia, Cuneo
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - I.R.S.T. Srl Irccs - Meldola - Sc Oncologia Medica, Meldola
  - Ao Ospedali Riuniti "Papardo Piemonte" - Po Papardo - Messina - Sc Ematologia, Messina
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Irccs Ospedale S. Raffaele - Milano - Unità Neoplasie Linfocitarie B, Milan
  - Aou Di Modena - Sc Ematologia, Modena
  - Aou Maggiore Della Carita' Di Novara - Scdu Ematologia, Novara
  - Aou Di Padova - Uo Ematologia, Padua
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagàni
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Ausl Della Romagna, Ospedale "Santa Maria Delle Croci" - Ravenna - Ematologia, Ravenna
  - Grande Ospedale Metropolitano "Bianchi-Melacrino-Morelli" Po E. Morelli - Reggio Calabria - Uoc Ematologia, Reggio Calabria
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Università degli Studi di Roma "Sapienza", Roma
  - Ao S. Maria - Terni - Sc Onco Ematologia, Terni
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Ospedale Mauriziano Umberto I - Torino - Scdu Ematologia, Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mauro FR, Starza ID, Messina M, Reda G, Trentin L, Coscia M, Sportoletti P, Orsucci L, Arena V, Casaluci GM, Marasca R, Murru R, Laurenti L, Ilariucci F, Stelitano C, Mannina D, Massaia M, Rigolin GM, Scarfo L, Marchetti M, Levato L, Tani M, Arcari A, Musuraca G, Deodato M, Galieni P, Patrizi VB, Gottardi D, Liberati AM, Giordano A, Molinari MC, Pietrasanta D, Mattiello V, Visentin A, Vitale C, Albano F, Neri A, De Novi LA, De Propris MS, Nanni M, Del Giudice I, Guarini A, Fazi P, Vignetti M, Piciocchi A, Cuneo A, Foa R. High rate of durable responses with undetectable minimal residual disease with front-line venetoclax and rituximab in young, fit patients with chronic lymphocytic leukemia and an adverse biological profile: results of the GIMEMA phase II LLC1518 - VERITAS study. Haematologica. 2023 Aug 1;108(8):2091-2100. doi: 10.3324/haematol.2022.282116. PMID 36632738
- See also: Gimema Foundation — http://www.gimema.it